CLINICAL TRIAL: NCT03780439
Title: Diagnostic Accuracy of Procalcitonin as an Early Predictor of Infection After Radical Gastrectomy for Gastric Cancer: a Prospective Bi-center Study
Brief Title: Procalcitonin to Predict Infection After Gastrectomy for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Yongchang Zhang (Other)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Yongchang Zhang, Hunan Province Tumor Hospital, Hunan Province Tumor Hospital
Organization: Hunan Province Tumor Hospital (Other)
Other Study IDs: PCT-INFECTION
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
Keywords: procalcitonin; infection; gastric cancer; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infection group and non-infection group: patients were divided into 2 sub-groups according to the presence of infection or not after radical gastrectomy for gastric cancer.

SUMMARY:
To investigate the diagnostic accuracy of procalcitonin as an early predictor of infection after radical gastrectomy for gastric cancer.

DETAILED DESCRIPTION:
From June 2018 to May 2019, consecutive eligible patients who underwent surgery for gastric cancer in the Department of Gastroduodenal and Pancreatic Surgery, Hunan Cancer Hospital and the treatment group of Professor Kai-xiong Tao in the Union Hospital of Tongji Medical College were invited to participate in the study. After surgery, routine blood test were measured morning on post-operative day (POD) 1, 3, 5, and 7, and serum level of procalcitonin was measured morning on POD 3 and 5.

The primary outcome of the present study was the accuracy of white blood cell (WBC) and neutrophil count, the neutrophil to WBC ratio (N%) and procalcitonin to detect post-operative infection (including intra-abdominal infection (IAI), surgical site infections (SSIs), pneumonia, urinary tract infection, catheter-related infection, and sepsis not specified) within 30 days after surgery. The main secondary outcome was their ability to detect any post-operative complications (such as intestinal obstruction, bleeding, ascites, cardiovascular and cerebrovascular events) within 30 days after surgery. Other secondary outcomes were the choice of the best timing to measure each inflammatory marker, the choice of a clinically meaningful cut-off value for the most accurate marker.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. pathologically diagnosed gastric adenocarcinoma
3. radical gastrectomy with lymphadenectomy.

Exclusion Criteria:

1. ongoing infection at surgery
2. pregnancy status
3. underwent non-resection surgery
4. underwent palliative gastrectomy
5. emergency surgery
6. taking corticosteroid or other immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pathologically diagnosed gastric adenocarcinoma who underwent radical gastrectomy.
Sampling Method: Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of procalcitonin to detect post-operative infection | within 30 days after surgery
  the accuracy of procalcitonin to detect post-operative infection

SECONDARY OUTCOMES:
diagnostic accuracy of procalcitonin to detect overall post-operative complications | within 30 days after surgery
  the accuracy of procalcitonin to detect any post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Hua Xiao, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Province Tumor Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Facy O, Paquette B, Orry D, Binquet C, Masson D, Bouvier A, Fournel I, Charles PE, Rat P, Ortega-Deballon P; IMACORS Study. Diagnostic Accuracy of Inflammatory Markers As Early Predictors of Infection After Elective Colorectal Surgery: Results From the IMACORS Study. Ann Surg. 2016 May;263(5):961-6. doi: 10.1097/SLA.0000000000001303. PMID 26135691
- [Result] Cousin F, Ortega-Deballon P, Bourredjem A, Doussot A, Giaccaglia V, Fournel I. Diagnostic Accuracy of Procalcitonin and C-reactive Protein for the Early Diagnosis of Intra-abdominal Infection After Elective Colorectal Surgery: A Meta-analysis. Ann Surg. 2016 Aug;264(2):252-6. doi: 10.1097/SLA.0000000000001545. PMID 27049766
- [Result] Xiao H, Quan H, Pan S, Yin B, Luo W, Huang G, Ouyang Y. Impact of peri-operative blood transfusion on post-operative infections after radical gastrectomy for gastric cancer: a propensity score matching analysis focusing on the timing, amount of transfusion and role of leukocyte depletion. J Cancer Res Clin Oncol. 2018 Jun;144(6):1143-1154. doi: 10.1007/s00432-018-2630-8. Epub 2018 Mar 23. PMID 29572591
- [Result] Munoz JL, Ruiz-Tovar J, Miranda E, Berrio DL, Moya P, Gutierrez M, Flores R, Pico C, Perez A. C-Reactive Protein and Procalcitonin as Early Markers of Septic Complications after Laparoscopic Sleeve Gastrectomy in Morbidly Obese Patients Within an Enhanced Recovery After Surgery Program. J Am Coll Surg. 2016 May;222(5):831-7. doi: 10.1016/j.jamcollsurg.2016.01.059. Epub 2016 Feb 13. PMID 27010585